CLINICAL TRIAL: NCT00002975
Title: A Phase II Trial of 4-5 Hour and 18-24 Hour Applications of 20% Topical ALA for Photodynamic Therapy of Cutaneous Carcinomas and Actinic Keratoses
Brief Title: Photodynamic Therapy in Treating Patients With Skin Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065494; RPCI-DS-96-55; NCI-G97-1224
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-08

CONDITIONS: Non-melanomatous Skin Cancer; Precancerous Condition
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin; actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Carcinoma, Basal Cell; Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDT (Experimental): 4-6h and 18-24h, 20%, ALA application of superficial and nodular epidermally-derived lesions using ca 633 nm laser irradiation
  Interventions: Drug: aminolevulinic acid

INTERVENTIONS:
Drug: aminolevulinic acid

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. Photodynamic therapy using aminolevulinic acid may be effective in treating patients with skin cancer.

PURPOSE: This randomized phase II trial is studying how well photodynamic therapy that includes aminolevulinic acid works in treating patients with skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of aminolevulinic acid and laser irradiation in patients with superficial and nodular epidermally derived lesions.

OUTLINE: This is a randomized study. Patients are stratified according to lesion type (superficial basal cell carcinoma [BCC] vs nodular BCC vs superficial squamous cell carcinoma vs actinic keratoses). Individual lesions on patients within each stratum are randomized to receive either a 4-5 or 18-24 hour application of aminolevulinic acid (ALA).

ALA is topically applied in a cream mixture and an occlusive dressing is placed over the lesion. After the randomized duration of ALA application has expired, the dressing is removed and a dye laser is used to treat the lesion.

Patients are followed for 2-5 years after treatment.

PROJECTED ACCRUAL: Up to 200 patients could be accrued, assuming 1 lesion per patient. 50 lesions are required for each stratified group.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Actinic keratoses
  * Histologically proven superficial or nodular basal cell carcinoma (BCC), squamous cell carcinoma in situ (Bowen's disease), or microinvasive squamous cell carcinoma
* No nodular BCC greater than 4 mm thick that will not be surgically removed
* No carcinoma with uncertain margins requiring Moh's surgery

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No known photosensitivity disease
* No porphyria or hypersensitivity to porphyrins

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior treatment with systemic photosensitizer that would cause residual cutaneous photosensitivity during study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 1997-02; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Zeitouni, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was activated in February, 1997, which was prior to Roswell Park Cancer Institute (RPCI) putting a system in place to centralize data entry and data management. Data entry was done by PI's staff. PI died and left incomplete data, and study was terminated in April, 2009.
Groups:
- Photodynamic Therapy Using 20% Topical ALA: 4-6h and 18-24h, 20%, ALA application of superficial and nodular epidermally-derived lesions using ca 633 nm laser irradiation
Period: Overall Study
Arm/Group | Photodynamic Therapy Using 20% Topical ALA
Started | 180
Treated With Study Therapy | 175
Completed | 175
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: Treated Patients
Arm/Group | Photodynamic Therapy Using 20% Topical ALA
Number analyzed (Participants) | 175
Age Continuous [Mean (Standard Deviation); unit: years] | 58.0 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 87

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Time Frame: One Year
Population: PI died, leaving incomplete data. Data not analyzed.
Arm/Group | Photodynamic Therapy Using 20% Topical ALA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: PI died, leaving incomplete data. No safety data from the trial were analyzed.
Arm/Group | Photodynamic Therapy Using 20% Topical ALA
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study was activated prior to RPCI putting a system in place to centralize data entry and data management. Data entry was done by PI's staff. PI died and left incomplete data. Efficay and safety data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes